CLINICAL TRIAL: NCT06278324
Title: Performance and Safety Assessment of HUMER STOP VIRUS Nasal Spray in Adults With Early Symptoms of Viral Respiratory Infection (COVID-19, Flu, Common Cold): an Open-label Randomized Controlled Study
Brief Title: Effectiveness of a Nasal Spray on Viral Respiratory Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: Urgo Research, Innovation & Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1736; 2023-A02286-39 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Tract Infection; Flu, Human; COVID-19; Common Cold
Keywords: Nasal spray
MeSH Terms: conditions — Influenza, Human; COVID-19; Common Cold

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, parallel arms (1:1 allocation ratio), single center, with a blind assessment for primary outcome
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of viral load analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal spray Humer Stop Virus (HSV) (Experimental): Patients treated with the nasal spray Humer Stop Virus (HSV) . Analgesics and antipyretics are authorized. Any other nasal spray, nasal cleansing (saline, water or other), and inhalation are prohibited
  Interventions: Device: Nasal Spray HSV Treatment
- Control (No Intervention): Analgesics and antipyretics are authorized. Any nasal spray, nasal cleansing (saline, water or other), and inhalation are prohibited

INTERVENTIONS:
Device: Nasal Spray HSV Treatment — Nasal treatment with the nasal spray Humer Stop Virus for 7 days, 2-3 puffs per nostril, 3-4 per day, space applications 4 hours apart.
  Arms: Nasal spray Humer Stop Virus (HSV)

SUMMARY:
There is no cure for cold or flu, most people recover in about within two weeks. Paracetamol may be used to reduce aches or treat fever, headache, or body aches. Antiviral solutions ranging from simple universal saline solutions to novel compounds have been proposed to provide a temporary barrier to prevent viral infection and propagation.

The nasal spray "Humer Stop Virus" is indicated in patients presented with early symptoms of viral respiratory infection. This spray forms a protective barrier in the nasal mucosa which is the main entry of the upper air respiratory system viruses. The spray traps the viruses and helps the organism to eliminate them before they multiply themselves.

This clinical investigation is conducted to assess the performance, clinical benefit and safety of this nasal spray in patients with early symptoms of acute respiratory disease whether or not infection is related to common cold, flu or COVID virus. Indeed, presence of early symptoms of acute respiratory infection does not always imply viral infectionAntigen self-tests are available to confirm viral infection with flu viruses or severe acute respiratory syndrome (SARS-CoV-2). However, influenza and other winter viruses are not systematically searched for in general population, because this is of neither collective nor individual interest. To be as pragmatic as possible, we chose to assess performance and safety of the nasal spray on intended users in real conditions. Patients with early symptoms of cold, flu or COVID, are enrolled regardless their PCR test positivity confirming viral infection at the time of enrollment. For study needs, the primary endpoint, which aims to assess the performance of the nasal spray in terms of stopping the viral infection, is assessed in a subgroup of patients with a positive PCR test with flu, COVID or common cold virus in the nasal sample collected at enrollment.

DETAILED DESCRIPTION:
Patients are recruited at the study site by the principal investigator, who gives a brief presentation of the study. Eligible, informed patients who sign a consent form are included and randomized.

All patients undergo three nasal swabs: at the time of enrolment, then 24 hours and 84 hours later, and complete a daily questionnaire on a secure mobile application dedicated to patient reported outcomes to assess their symptoms and provide information on any analgesic or antipyretic medication they may have been taking.

Patients randomized to the intervention group are asked to use the nasal spray as recommended and to report any difficulties with the device.

A final visit is organized on day 8 at the investigation center under the supervision of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* With early symptoms of respiratory infection (onset less than 48 hours before inclusion) of mild to moderate intensity (TSS ≥ 2 and < 9).
* Having a mobile phone allowing using the patient reported outcome App. (NursTrial®).
* Patient able to understand and comply with protocol requirements and instructions, including answering a questionnaire on a mobile phone, as required by protocol.
* Signed informed consent.
* Affiliated to a French Health insurance scheme.

Exclusion Criteria:

* Concomitant disease or infection that could interfere with participation in the study: acute ear, nose, and throat and respiratory tract disease other than the common cold, flu or COVID (e.g., tonsillitis, otitis, bronchitis) and chronic sinusitis or allergic rhinitis, or other reasons for nasal obstruction and other past or present conditions and treatments that could influence symptom scores.
* Severe nasal septum deviation or other conditions that could cause nasal obstruction such as the presence of nasal polyps.
* Known or suspected intolerance or hypersensitivity, including history of allergies, to any component investigational device material, any history of drug hypersensitivity.
* Concomitant treatment that might impair the trial results (i.e., decongestants, local anesthetics, topical corticosteroids, saline solution) during the seven days prior to inclusion.
* Smokers.
* Have a condition or is taking a medication that the Investigator and/or designee believes could jeopardize the safety of the subject, would interfere with the evaluation, or confound the interpretation of the study results.
* Non-compliant or may not respect the constraints imposed by the protocol.
* Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial;
* Woman of childbearing age (except menopausal, hysterectomised, sterilized) not using effective contraception (oral contraceptives, intra-uterine device, contraceptive implant, or condoms).
* Person belonging to a population referred to in articles 64 (incapacitated subjects), 65 (minors), 66 (pregnant or breastfeeding women), 67 (persons performing mandatory military service, persons deprived of liberty, persons who, due to a judicial decision) and 68 (patients in emergency) of the Medical Device Regulation.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Performance of nasal spray in eliminating viruses | 84 hours
  0-84 hours areas under the curve (AUC) of viral load in patients with a positive virus infection at enrollment.
  Positive viral infection means that at least one of the following respiratory viruses has been detected in nasal sample collected at enrollment: SARS-CoV-2, Influenza A virus, Influenza B virus, Respiratory syncytial virus (RSV) A/B, Metapneumovirus (MPV), Adenovirus A/B/C/D/E/F, Rhinovirus A/B/C, Parainfluenza virus 1/2/3/4, Bocavirus 1/2/3/4, Coronavirus 229E, Coronavirus NL63, Coronavirus OC43 Virus load is measured using Reverse Transcriptase quantitative polymerase chain reaction (RT-qPCR).

SECONDARY OUTCOMES:
Changes from baseline in viral load | 24 hours and 84 hours
  Percentage reduction in viral load in patients with a positive virus infection at enrollment.
  Virus load is measured as described in primary outcome.
Rate of patients cleared from viral infection | 24 hours and 84 hours
  Percentage of patients with a positive virus infection at enrollment totally cleared from viral infection, meaning with negative viral load.
  Virus load is measured as described in primary outcome.
Rate of patients with improved viral infection | 24 hours and 84 hours
  Percentage of patients with a positive virus infection at enrollment who present lower viral load.
  Virus load is measured as described in primary outcome.
Rate of patients with worsening viral infection | 24 hours and 84 hours
  Percentage of patients with a positive virus infection at enrollment who present higher viral load.
  Virus load is measured as described in primary outcome.
Rate of patients with new viral infection | 24 hours and 84 hours
  Percentage of patients with a virus infection not present at enrollment. Virus load is measured as described in primary outcome.
Changes in symptom severity | day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Symptom severity is assessed using the Total Symptom Score, which consists of 7 questions, each rated on a 4 point-Likert scale (none = 0, mild = 1, moderate = 2, severe = 3).
  The score ranges from 0 to 28.
Duration of illness | day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Number of days between onset of symptoms and last day before first day with Total Symptom Score returns to 0.
  Total Symptom Score is measured as described in outcome 7
Time to clinical improvement of the symptoms | day 1, day 2, day 3, day 4, day 5, day 6, day 7
  Number of days between day 1 and the first day the patient reports "much improved" or "very much improved," items of the 7 point-Likert scale assessing the patient's global impression of improvement
Adverse event occurence | day 8
  Percentage of patients with adverse events between consent signature and final visit.

OTHER OUTCOMES:
Patient opinion of nasal spray | day 8
  Patients treated with the nasal spray complete a satisfaction questionnaire designed for the study, and their responses are assessed using Likert scales.
Nasal spray safety | Day 8
  Frequency and description of device deficiencies or difficulties in using the nasal spray reported by patients treated with the nasal spray.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle FOUCHER, Study Director — Urgo Research, Innovation & Development
Locations (1):
- Cen Experimental, Dijon, Burgundy, France

IPD SHARING:
Plan to Share IPD: No